CLINICAL TRIAL: NCT02670174
Title: Influence of Kinetic Chain Training on the Treatment Outcome of Overhead Athletes With Shoulder Impingement Syndrome
Brief Title: Influence of Kinetic Chain Training on the Treatment Outcome of Overhead Athletes With Impingement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015/0816
Record Dates: First submitted 2015-09-29; First posted 2016-02-01 (Estimated); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Shoulder Impingement Syndrome
Keywords: Shoulder impingement syndrome; Overhead athletes; Kinetic chain; Exercise treatment
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Intervention Model Description: Subjects are randomly assigned in 3 parallel intervention groups. They cannot participate in 2 or more intervention groups.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Traditional training (Active Comparator): A home exercise program consisting of rotator cuff and scapular muscle training will be performed during 6 weeks (4 sessions/week). To monitor progress and control load progression, a physical therapist will visit the subject every week.
  Interventions: Other: Traditional training
- Separate kinetic chain training (Experimental): A home exercise program consisting of traditional training exercises as well as separate exercises focusing on core and lower limb training will be performed during 6 weeks (4 sessions/week). To monitor progress and control load progression, a physical therapist will visit the subject every week.
  Interventions: Other: Separate kinetic chain training
- Integrated kinetic chain training (Experimental): A home exercise program consisting of traditional training exercises while integrating core and lower limb training will be performed during 6 weeks (4 sessions/week). To monitor progress and control load progression, a physical therapist will visit the subject every week.
  Interventions: Other: Integrated kinetic chain training

INTERVENTIONS:
Other: Traditional training
  Arms: Traditional training
Other: Separate kinetic chain training
  Arms: Separate kinetic chain training
Other: Integrated kinetic chain training
  Arms: Integrated kinetic chain training

SUMMARY:
A randomized controlled trial will be conducted to examine the effectiveness of a traditional home exercise program versus 2 kinetic chain home exercise programs on treatment outcome of overhead athletes with shoulder impingement syndrome. Primary outcome measures are reduction of pain and disability, and improvement in functionality and sports performance. Secondary outcome measures are strength, mobility, flexibility and functional performance.

DETAILED DESCRIPTION:
Participant are randomly assigned in 3 home exercise groups.

1. The traditional program: consists of solely strengthening the rotator cuff muscles and scapular muscles (e.g. external rotation)
2. Separate kinetic chain program: same exercises as the first group but they also receive an exercise program to separately train the core and lower body. (e.g. external rotation separately and squat separately)
3. Integrated kinetic chain program: same exercises as the first group but all exercises are performed while simultaneously activating the kinetic chain. (e.g. external rotation while squatting).

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of shoulder impingement on the dominant side for at least 3 months and at least 3 of the following tests are considered positive

  * Jobe
  * Hawkins
  * Neer
  * Painful arc during elevation
  * Pain or lack of force production with isometric external rotation
  * Apprehension test
  * Relocation test
* Performing overhead sports at least 3 hours/week
* Shoulder pain interferes with sports activities
* They have not had treatment for this shoulder pain

Exclusion Criteria:

* History of shoulder dislocation or subluxation
* History of orthopedic surgery
* No complaints of pain or dysfunction in the upper limb (except impingement related complaints in the dominant shoulder), lower limb or spine at the last 6 months
* Currently taking nonsteroidal anti-inflammatory medication
* Received a steroid injection in the past 12 months
* Participating in another study
* Known systemic diseases
* Known structural diseases

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2015-09; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Changes in Shoulder Pain And Disability Index (SPADI) score | At baseline and within one week after the 6-weeks training program
  Patients will fill in the SPADI questionnaire to evaluate shoulder pain and function. The SPADI is a valid, reliable and frequently used questionnaire for shoulder pain patients consisting of 13 items divided in 2 subscales: pain (5 items) and disability (8 items). Each item was scored on a 10-point numeric rating scale. Total and subscale scores were summed and transformed to a score out of 100 (%) were a higher score indicates a higher level of pain and/or disability
Changes in Western Ontario Shoulder Stability index (WOSI) score | At baseline and within one week after the 6-weeks training program
  The WOSI is a patient-evaluated disease-specific quality of life scoring questionnaire that has been developed for shoulder instability patients. This 21-item questionnaire consists of 4 subscales: physical symptoms (10 items), sport/recreation/work (4 items), lifestyle (4 items), and emotions (3 items). Each item was scored on a 100-mm visual analogue scale. Total and subscale scores were summed and transformed to a score out of 100 (%) where a higher score indicates more limitations in shoulder related quality of life
Subjective perception of shoulder improvement | 6-weeks training program
  A Global Rating of Change (GROC) scale was used to quantify patient-perceived improvement of overall shoulder function after 6 weeks treatment as "improved", "unchanged" or "worse". In case they improved or got worse, the amount of change was reflected on a 5-point scale: very little change, little change, some change, a large change, a very large change. An "unchanged" condition scored 0, "improved" between 1 and 5, and "worse" between -1 and -5 points.
  amount of change was scored on a 5-point scale (very little change, little change, some change, a large change, a very large change)

SECONDARY OUTCOMES:
Changes in shoulder muscle isokinetic strength (Biodex system 4) | at baseline and within one week after the 6-weeks training program
  Isokinetic strength of shoulder internal and external rotators will be measured bilateral with the Biodex device (Biodex system 4, Biodex Medical Systems, Inc., Shirley, New York, USA). For further analysis, concentric peak torque (PT) (rotation) or peak force (PF) (protraction-retraction) values were normalized to body weight (BW). A higher value represents more strength and thus a better outcome.
Changes in shoulder scapular isokinetic strength | at baseline and within one week after the 6-weeks training program
  Isokinetic strength of scapular protraction and retraction muscles will be measured bilateral with the Biodex device (Biodex system 4, Biodex Medical Systems, Inc., Shirley, New York, USA). For further analysis, concentric peak torque (PT) (rotation) or peak force (PF) (protraction-retraction) values were normalized to body weight (BW). A higher value represents more strength and thus a better outcome.
Changes in scapular dyskinesis | at baseline and within one week after the 6-weeks training program
  Scapular dyskinesis will be measured by observing the scapular movement during active elevation. For both sides (left and right), scapular dyskinesis was evaluated as being present or not. In case dyskinesis was present, the amount of dyskinesis is scored as subtle or prominent.
Changes in functional tests for the upper limb measured with the Y Balance Test | at baseline and within one week after the 6-weeks training program
  The YBT-UQ is a commonly used upper extremity functional test to assess closed kinetic chain function of the stance arm while performing an open kinetic chain movement in the reaching arm. Under standardized verbal encouragement, patients stand in a three point plank position while using the free arm to push a reach indicator box as far as possible in 3 reach directions i.e. medial, inferolateral and superolateral.The average of the 3 test trials for each limb and each direction was normalized for upper limb length. Additionally, a normalized composite score per side was calculated by averaging the mean normalized test scores in the 3 reach directions. A higher scores indicates a better outcome.
Return To Play (RTP) | up to one week after the 6-weeks training program
  Is it possible to return to play after 6 weeks intervention or not? In addition, following question was asked: on a scale of 0 to 100%, what is the extent to which the injured shoulder has reached the shoulder function before the injury occurred?
Changes in functional tests for the upper limb measured with the Seated Medicine Ball Throw | at baseline and within one week after the 6-weeks training program
  The SMBT is an open kinetic chain functional screening test to assess bilateral upper body power and strength. The subjects were instructed to sit on the floor with the head, shoulder and back against the wall while holding a 2kg medicine ball with both arms.Participants had to throw the medicine ball forward, in a straight line and as far as possible with head, shoulders and back maintaining full wall contact. For further analysis, the mean distance of 4 test trials was calculated. A higher scores indicates a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Cools, PT, PhD, Principal Investigator — University Ghent
Locations (1):
- Vakgroep REVAKI (Ghent University - Ghent University hospital), Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No